CLINICAL TRIAL: NCT02226861
Title: Ultra Low Dose IL-2 Therapy as GVHD Prophylaxis in Haploidentical Allogeneic Stem Cell Transplantation
Brief Title: Ultra-Low Dose IL-2 Therapy as GVHD Prophylaxis in Haploidentical Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 140180; 14-H-0180
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-06-27

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Chronic Lymphocytic Leukemia (CLL); Chronic Myelogenous Leukemia (CML); MDS
Keywords: Acute Lymphoblastic Leukemia (ALL); MDS; Chronic Myelogenous Leukemia (CML); Chronic Lymphocytic Leukemia (CLL); Acute Myelogenous Leukemia (AML)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

ARMS (1):
- 1 (Experimental): Subjects will receive CD34-selected stem cells followed by fixed dose ULG IL-2 (100,000 IU/m2) given subcutaneously for 12 weeks+Sirolimus until Day +60
  Interventions: Device: CliniMACS CD34 selection system; Biological: ULD IL-2

INTERVENTIONS:
Device: CliniMACS CD34 selection system — Stem cells will be selected with the CliniMACS system before transplant.
Biological: ULD IL-2 — sterile, white to off-white, preservative-free, lyophilized powder suitable for IV infusion upon reconstitution and dilution

SUMMARY:
Background:

- Stem cell transplantation from a partially matched donor can lead to graft-versus-host disease (GVHD). Researchers want to learn how to improve these transplantations.

Objective:

- To see if very low doses of Interleukin-2 after a partially matched transplantation prevent GVHD.

Eligibility:

* Recipients: age 18 65, with certain bone marrow or lymphatic system diseases and an available family member with partial tissue match.
* Donors: age 18 80.

Design:

* Recipients will be screened with medical history, physical exam, and many tests including blood and tissue tying.
* Donors will be screened with medical history, physical exam, blood tests and tissue typing.
* Recipients will stay in the hospital 3 6 weeks.
* All participants will have apheresis. Blood is drawn from one arm, run through a machine that collects white blood cells, then returned into the other arm.
* Recipients will have:
* Intravenous (IV) line placed under the skin and into a neck vein, to stay throughout transplant and recovery. They may also have a catheter inserted for collecting immune cells.
* Bone marrow sample taken by needle. They will have 3 more after transplant.
* Donors will have:
* Filgrastim injected once daily for 5 6 days.
* Stem and immune cells collected by another apheresis.
* Recipients will get:
* Eight 30-minute doses of radiation, sitting at a machine.
* Donor immune cells by IV, 6 days before the transplant day.
* Chemotherapy drugs by IV.

<TAB><TAB>- Donor stem cells by IV on transplant day.

* After transplant, recipients will give self-injections of very low doses of Interleukin-2 once daily for about 12 weeks.
* Before and after transplant, recipients will get medicine to suppress the immune system and antibiotics to prevent infections
* Recipients must stay near NIH for 3 6 months after transplant.
* All recipients and donors will have 3 years of follow-up.

DETAILED DESCRIPTION:
Although allogeneic stem cell transplantation (allo-SCT) is a curative option for many hematologic malignancies, not all have a suitable donor. Haploidentical peripheral blood stem cell transplantation (haplo-SCT) has the advantage of immediate availability, higher stem cell dose, and feasibility of repeated cell collections for generating lymphocyte infusions to treat or prevent relapse or infection. However, haplo-SCT incurs a risk of bidirectional rejection with either severe graft versus host disease (GVHD) or graft rejection by the recipient. Therefore it is important to develop novel strategies to optimize the outcome of haplo-SCT. Designing a haplo-SCT that incorporates the concepts of modulating the immune system and allowing the opportunity for graft manipulation and/or adoptive immunotherapy may improve the treatment outcome. To achieve this, we are first interested in studying the immune modulatory effect of ultra-low dose Interleukin 2 (ULD IL-2) as GVHD prophylaxis.

This is an investigator initiated pilot study to determine the safety and feasibility of ULD IL-2 as GVHD prophylaxis in haploidentical allogeneic stem cell transplantation for patients with hematologic malignancies. Because GVHD has previously been associated with low numbers of circulating CD4+ CD25+FOXP3+ regulatory T cells (T(regs)), research efforts in increasing T(regs) either ex-vivo with adoptive transfer of T(regs) or in vivo using immunomodulatory agents such as IL-2, have shown promise in reducing incidences of GVHD.

The primary objective of this study is to evaluate safety and feasibility. Secondary objectives are to determine the incidences of acute and chronic GVHD, engraftment, overall survival, transplant related mortality, and relapse.

We will adopt the 2 step haplo-SCT method developed by Grosso et. al1 to study our method of GVHD prophylaxis. This 2 step approach, in which the lymphoid and myeloid portions of the graft are given in two separate steps in order to control and optimize T-cell, has already been published as a feasible and safe platform for haplo SCT for patients with hematologic malignancies and has been adopted by the Jefferson University Hospital (PA, USA), where they continue to treat patients under this protocol. As an additional GVHD prophylaxis, we will use sirolimus, an previously established GVHD prophylaxis which may work with ULD IL-2 synergistically to increase T(regs) .

The haploidentical donor will be mobilized by G-CSF and undergo one apheresis to collect lymphocytes and CD34+ stem cell product after Miltenyi CD34+ selection. The products will be cryopreserved until the time of transplantation. Recipients will receive a myeloablative conditioning regimen of fludarabine and total body irradiation (TBI) on days -10 to -6. After the last fraction of TBI, a donor lymphocyte infusion (DLI) product (2 times 10(8) CD3+/kg) will be given. Cyclophosphamide will be given on days -3 and -2, followed by CD 34+ selected donor stem cell product infused on day 0. Sirolimus will be initiated on day -1 until day+60. ULD-IL2 (100,000 IU/m2) will give subcutaneously daily for 12 weeks starting day +1.

This study will evaluate 14 recipients (ages greater than or equal to 18 - less than or equal to 75; planned accrual up to 20 recipient in event of replacement) with hematologic malignancies meeting indication for transplant but who do not have matched related or unrelated donor available. Safety will be monitored continuously with a stopping rule for toxicity based on the treatment-related serious adverse event rate (TRSAE). Safety monitoring will continue until at least 114 days after transplantation, and recipients experiencing adverse events will be monitored until toxicity resolution or stabilization. Stopping rule is defined as nonrelapse mortality and steroid refractory GVHD during the period of safety monitoring for ULD IL-2. Recipients will be followed for up to 1 year to evaluate the incidences of acute and chronic GVHD, engraftment, overall survival, transplant related mortality, and relapse.

ELIGIBILITY:
* INCLUSION CRITERIA RECIPIENT:
* Ages 18-70 years inclusive
* Haploidentical donor available
* Any one of the following hematologic conditions meeting a standard indication for allogeneic stem cell transplant:

  * Chronic myelogenous leukemia (CML): Subjects under the age of 21 in chronic phase OR subjects ages 18-65 in chronic phase who have failed treatment with imatinib or have intolerance to imatinib OR Subjects ages 18-65 in accelerated phase or blast transformation. OR
  * Acute lymphoblastic leukemia (ALL): any of these categories: Adult ALL including standard risk. All second or subsequent remissions, primary induction failure, partially responding or untreated relapse. OR
  * Acute myelogenous leukemia (AML): AML in first remission - except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), c-kit unmutated AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse. OR
  * Myelodysplasticsyndromes(MDS): any of these categories - refractory anemia with transfusion dependence, refractory anemia with ANC<500/ (Micro)L, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia, atypical MDS/myeloproliferative syndromes. OR
  * Myeloproliferative disorders including atypical (Ph-negative) chronic myeloid and neutrophilic leukemias, progressing myelofibrosis, and polycythemia vera, essential thrombocythemia either in transformation to acute leukemia or with progressive transfusion requirements or pancytopenia. OR
  * Non-Hodgkin s lymphoma including Mantle cell lymphoma relapsing or refractory to standard of care treatments. OR
  * Multiple myeloma, Waldenstroms macroglobulinemia, unresponsive or relapsed following standard of care treatments. OR
  * Hodgkin's Lymphoma relapsing following an autologous transplant. OR
  * Other rare hematologic malignancies for which hematopoietic stem cell transplantation has been performed and offers a durable remission or as the only option with a potential for cure.

    * Chemotherapy-resistant multisystem Langerhans cell histiocytosis (MSLCH) especially involving organs like the bone marrow, liver, spleen, and lungs
    * Aggressive systemic mastocytosis, and mast cell leukemia (MCL) in first CR (CR1)
    * Hypereosinophilic syndrome who have failed imatinib therapy or FIP1L1-PDGFRa-negative patients who develop end-organ dysfunction
    * Adult T-cell leukemia/lymphoma at first diagnosis
    * Refractory or disseminated nasal-type extranodal NK/T-lymphoma or aggressive Natural killer cell leukemia/lymphoma
    * Mycosis fungoides and S(SqrRoot)(Copyright)zary syndrome after failure of two or three initial therapies
    * Primary or relapsed refractory Angioimmunoblastic T-cell lymphoma at first diagnosis
    * Hepatosplenic T-cell lymphoma (gamma/delta T-cell lymphoma) at first diagnosis
    * T-cell prolymphocytic leukemia at first diagnosis
    * Subcutaneous panniculitic T-cell lymphoma at first diagnosis
    * Hematodermic neoplasm (blastic natural killer cell lymphoma or Blastic plasmacytoid dendritic cell neoplasm) at first diagnosis
  * Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA RECIPIENT (ANY OF THE FOLLOWING):

* HLA identical (6/6) related or (8/8 allele level matched) unrelated donor available and readily accessible at time of transplantation evaluation
* Major anticipated illness or organ failure incompatible with survival from transplant
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and making informed consent impossible.
* Positive pregnancy test for women of childbearing age
* Contraindication to receive IL-2 including:

  * Hypersensitivity to IL-2
  * Sustained ventricular tachycardia (>5 beats)
  * Cardiac arrhythmias not controlled or unresponsive to management
  * Chest pain with ECG changes, consistent with angina or myocardial infarction
  * Cardiac tamponade
  * Intubation for >72 hours
  * Renal failure requiring dialysis >72 hours
  * Coma or toxic psychosis lasting > 48 hours
  * Repetitive or difficult to control seizures
  * Active bowel ischemia or perforation
  * Active GI bleeding requiring surgery
* DLCO adjusted for Hb and ventilation< 50% predicted
* Left ventricular ejection fraction < 40% (evaluated by ECHO) or < 30% (evaluated by MUGA)
* AST/SGOT > 5 times ULN
* Total bilirubin > 3 times ULN
* Estimated GFR <60ml/min (calculated by CKD-EPI, a formula routinely used in Clinical Research Center at National Institutes of Health. In case of borderline estimated GFR, CKD-EPI creatinine-cystatin C formula will be used for more accurate estimation)
* Prior allogeneic stem cell transplantation

INCLUSION CRITERIA DONOR:

* Related donor who shares 1 haplotype with the recipient
* Age greater than or equal to 18 or less than or equal to 80 years old
* Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA DONOR (ANY OF THE FOLLOWING):

* Unfit to receive G-CSF and undergo apheresis such as abnormal blood counts, history of stroke, uncontrolled hypertension
* Sickling hemaglobinopathy including HbSS, HbAS, HbSC
* Donors who are positive for HIV, active hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II)
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08-26; Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Safety of ULD IL-2 as GVHD proph | 4 months
  The primary endpoint to this study is to evaluate the safety of ULD IL-2 as GVHD prophylaxis in haploidentical transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Sawa Ito, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grosso D, Carabasi M, Filicko-O'Hara J, Kasner M, Wagner JL, Colombe B, Cornett Farley P, O'Hara W, Flomenberg P, Werner-Wasik M, Brunner J, Mookerjee B, Hyslop T, Weiss M, Flomenberg N. A 2-step approach to myeloablative haploidentical stem cell transplantation: a phase 1/2 trial performed with optimized T-cell dosing. Blood. 2011 Oct 27;118(17):4732-9. doi: 10.1182/blood-2011-07-365338. Epub 2011 Aug 25. PMID 21868572
- [Background] Barrett J, Gluckman E, Handgretinger R, Madrigal A. Point-counterpoint: haploidentical family donors versus cord blood transplantation. Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S89-93. doi: 10.1016/j.bbmt.2010.10.024. No abstract available. PMID 21195317
- [Background] Fuchs EJ. Haploidentical transplantation for hematologic malignancies: where do we stand? Hematology Am Soc Hematol Educ Program. 2012;2012:230-6. doi: 10.1182/asheducation-2012.1.230. PMID 23233586